CLINICAL TRIAL: NCT02525406
Title: Models for Improving Operating Room Productivity: Delays, Cancellations and Pre-admission Testing
Status: Active, not recruiting | Type: Observational
Sponsor: University of Toledo Health Science Campus (Other)
Responsible Party: Sponsor
Organization: University of Toledo (Other)
Other Study IDs: Surgical-Cancellation-Study
Record Dates: First submitted 2015-07-21; First posted 2015-08-17 (Estimated); Last update posted 2025-06-27 (Actual); Status verified 2025-04

CONDITIONS: Other Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: All surgeries performed from Jan 01, 2010 to Aug 31, 2020

SUMMARY:
The goal of the study is to identify factors that enhance productivity and increase value delivered by hospitals drawing on concepts used in industry for quality and productivity in production and operations management literature. The investigators intend to look at surgeon experience, patient characteristics and pre-admission testing on operating room productivity.

ELIGIBILITY:
Inclusion Criteria:

* All scheduled surgical patients' information gathered in Surgery database from January 2010 thru August 2020 will be included.

Exclusion Criteria:

* Any case type where less than 5 surgeries were performed by a surgeon would be excluded and if the surgeon in question had less than 3 months of data available.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients scheduled for surgery at UTMC from Jan 01,2010 to August 31, 2020
Sampling Method: Probability Sample
Enrollment: 9240 (Estimated)
Dates: Start 2015-07; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Surgical Experience vs Average Completion times of surgical procedures | intraoperative
  A measurement of the surgeon's experience (in years) since completion of training until the surgical procedure (Day of surgery/Day 1) will be compared to the surgeon's average time (measured in minutes) to complete the surgical procedure.

SECONDARY OUTCOMES:
Variability in Completion times of surgical procedures to predict scheduling difficulties. | intraoperative
  The length of time (measured in minutes) required to complete surgical procedures will be assessed for variability per surgeon. Extreme variability will be compared to the effect on the surgery schedule for that date.
Preadmission Testing and how it relates to the surgical procedure: time to completion, delays in starting time and/or cancellation. | Day 1
  Patients completing testing and assessment in the Pre Admission testing center will be compared to patients that were not tested or assessed in the Pre admission testing center to determine if there is a change in the completion time of the surgical procedure, increase the variability in the completion time for the surgeon, lead to delays or cancellation of the surgical procedures.
Patient Acuity vs Complexity of surgical procedure | Day 1
  The patient acuity level will be compared to the complexity of the surgical procedure as measured by an investigator assigned complexity scale and how it relates to the time to completion and its impact on operating room scheduling.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew B. Casabianca, MD, Principal Investigator — University of Toledo
Locations (1):
- University of Toledo, Toledo, Ohio, United States